CLINICAL TRIAL: NCT03079570
Title: A Pilot Study Examining Differences in Critical Flicker Fusion Thresholds Between Young and Old Subjects With Normal Ocular Health at Photopic, Mesopic, and Scotopic Luminance Levels
Brief Title: Flicker Fusion Thresholds Between Young and Old Subjects at Various Luminance Levels
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-270-0007
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Age Factor; Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to determine which luminance levels yield maximum differences in critical flicker fusion (CFF) scores between younger and older normal subjects.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a chronic, progressive eye disease. AMD is one of the leading causes of visual impairment and blindness among elderly populations in economically developed countries . Due to the aging of the population, the incidence and prevalence of AMD is likely to increase substantially over the next decade, potentially posing a significant impact on society.

AMD is a complex and progressive degenerative disease, with both genetic and environmental risk factors. AMD affects the outer retina, retinal pigment epithelium (RPE), Bruch's membrane, and choroid. The retina is among the most metabolically active tissues in the body, in part due to rods, which frequently discard their outer segments tips, and the RPE, which phagocytoses the discarded tips . The retina's metabolism causes accumulation of toxic by-product by the following: 1. Energy metabolism (oxidative stress); 2. Visual cycle modulator (lipofuscin); 3. Local inflammation (complement activation). The local inflammation, and the accumulation of lipofuscin material within the RPE, may lead to drusen formation, RPE dysfunction, and degeneration of macular rods and cones, finally leading to the irreversible loss of vision.

AMD occurs in two forms - a non-exudative "dry" form and an exudative "wet" form. Non-exudative AMD accounts for 80-90% of AMD cases and it involves a diverse phenotype that may include drusen and/or RPE pigmentation abnormalities. Advanced non-exudative AMD is characterized by geographic atrophy, which is characterized by the presence of an expanding region of irreversible RPE and photoreceptor loss in the macula.

At the present time, there are no approved treatments for non-exudative AMD. The clinical development of therapeutic agents for the treatment of non-exudative AMD is limited by slow disease progression, unsuitability of commonly used efficacy endpoints such as visual acuity, and difficulty in identifying those subjects with early stages of disease most likely to progress. Visual function testing may prove to be useful tools in detecting the early non-exudative AMD.

In early age-related macular degeneration, outer retinal metabolism is known to be compromised. The detection of a flickering stimulus imposes a higher metabolic requirement than does a static stimulus , . Inability to detect a flickering stimuli may identify earlier stages of disease than the inability to detect static stimuli. Early work by Mayer, et.al. has shown that AMD subjects experience functional deficits in the mid range of visual phenomenon most notably at 10HZ and 14Hz. Phipps, et.al. found early AMD subjects to have larger deficits for flickering than static stimuli . Later work has shown that a flicker test based on mid-range frequencies has been shown to have effective diagnostic and reproducibility characteristics relative to other functional tests . In addition to the diagnostic potential of flicker stimuli, this test has been shown to be predictive of AMD progression and correlated to AMD severity . Therefore, a flicker test may prove useful in identifying early dysfunction in macular performance and for assessment treatment in future interventional clinical trials.

Critical Flicker Fusion (CFF) is a type of flicker test that involves increasing the frequency of a flashing stimulus until that stimulus appears static to an observer. The frequency at which critical flicker fusion occurs is recorded as a patient specific endpoint of visual function. In this study, we will investigate CFF across a wide range of luminance levels, from photopic to scotopic ranges, in young and old subjects with normal ocular health. The impact of age on CFF threshold will be the focus of this study, with the primary objective being to highlight luminance levels where maximum differences between young and old subjects occur.

ELIGIBILITY:
Inclusion Criteria:

* Provide written and informed consent;
* Be willing and able to follow all instructions and attend the study visit;
* Must be able to successfully complete all study procedures;
* If female and of childbearing potential, not be pregnant, nursing, or planning a pregnancy and be willing to submit a pregnancy test at Visit 1 (and exit visit as applicable) and utilize an acceptable form of birth control for the duration of the study;
* Be 18 years of age or older
* Have best-corrected distance visual acuity (BCVA) of better or equal to 20/30 in at least one eye at Visit 1;
* Have best-corrected near visual acuity of better or equal to 20/30 in at least one eye at Visit 1;
* Have visited an ophthalmologist for an eye exam within 1 year of Visit 1;

Exclusion Criteria:

* Have a history of age-related macular degeneration (exudative and non-exudative), diabetic retinopathy, retinal detachment, or any chronic retinopathy or retinal degenerative disease;
* Have had prior retinal vein or artery occlusion, history of macular edema, or optic neuropathy;
* Have a history of glaucoma or ocular hypertension
* Have visually significant cataracts at Visit 1;
* Have a history of ocular trauma;
* Have a history of photophobia reported at Visit 1;
* Report ocular discomfort of 2 or greater in either eye at Visit 1, or report any other ocular symptomatology that could in the opinion of the investigator interfere with study procedures;
* Have active signs or symptoms of conjunctivitis, uveitis, in either eye at the baseline examination of Visit 1;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 7 days of entry into this study;
* Have used contact lenses 24 hours prior to the start of the study or be unwilling to discontinue wearing for the duration of the study;
* Have a history of uncontrolled systemic disease (e.g. poorly controlled hypertension or poorly controlled diabetes, a history of status asthmaticus, organ transplant) at Visit 1;
* Have a history of seizures;
* Be currently taking procyclidine, alprazolam (Xanax), lorazepam (Ativan), Adderall, or any psychotropic medications;
* Be a woman who is pregnant or nursing an infant
* Have a condition or be in a situation that the investigator feels may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects at least 18 years of age with healthy eyes and good vision
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
Mean Critical Flicker Fusion Scores | At each luminance level (about 5 minutes between each)
  Critical flicker fusion threshold (Hz) will be measured at each designated luminance level
Percentage Difference Between Population | At each luminance level (about 5 minutes between each)
  Critical flicker fusion scores between populations will be compared at luminance levels

SECONDARY OUTCOMES:
Percent Change | At each luminance level (about 5 minutes between each)
  Mean percent change of critical flicker fusion scores between luminance levels

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Chin, OD, Principal Investigator — Practicing Physician
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No